CLINICAL TRIAL: NCT05492201
Title: A Single Ascending and Multiple Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3873862 in Healthy Participants
Brief Title: A Study of LY3873862 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18445; J3X-MC-LYGA (Other: Eli Lilly and Company); 2022-000500-36 (EudraCT Number)
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- LY3873862 (Part A) (Experimental): LY3873862 administered orally as single dose.
  Interventions: Drug: LY3873862
- Placebo (Part A) (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo
- LY3873862 (Part B) (Experimental): LY3873862 administered orally as multiple doses.
  Interventions: Drug: LY3873862
- Placebo (Part B) (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo
- LY3873862 (Part C) (Experimental): LY3873862 administered orally as multiple doses.
  Interventions: Drug: LY3873862
- Placebo (Part C) (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3873862 — Administered orally.
  Arms: LY3873862 (Part A); LY3873862 (Part B); LY3873862 (Part C)
Drug: Placebo — Administered orally.
  Arms: Placebo (Part A); Placebo (Part B); Placebo (Part C)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3873862 when administered either in single or multiple doses in healthy participants. The study will also assess how fast LY3873862 gets into the blood stream and how long it takes the body to remove it. The study is open to healthy participants. The study will last up to approximately 58, 72, and 72 days for Part A, B, and C, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation
* Body mass index (BMI) within the range 18.0 to 32.0 kilograms per meter squared (kg/m²)
* Are male or female participants, including those of childbearing potential

Exclusion Criteria:

* Have a history or presence of medical illness including, but not limited to, any cardiovascular, renal, hepatic, gastrointestinal, respiratory, hematologic, endocrine, psychiatric, or neurological disease, convulsions, or any clinically significant laboratory abnormality that, in the judgment of the investigator, indicate a medical problem that would preclude study participation.
* Are unwilling to comply with the dietary restrictions required for this study, including the avoidance by 5 days prior to study drug administration until the final ambulatory visit the ingestion of fruits, sauces, and juices containing furanocoumarins that irreversibly inhibit cytochrome P450 (CYP)3A4. The following fruits, sauces, and juices are excluded: grapefruit, Seville oranges, pomelos, cranberry, Goji berry, and apple.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through 72 days
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of LY3873862 | Predose up to 96 hours postdose
  PK: AUC[0-∞] of LY3873862
PK: Area Under the Concentration versus Time Curve at Steady State (AUCτ) of LY3873862 | Predose up to 96 hours postdose
  PK: (AUCτ) of LY3873862
PK: Maximum Observed Concentration (Cmax) of LY3873862 | Predose up to 96 hours postdose
  PK: Cmax of LY3873862
PK: Time of Maximum observed Concentration (Tmax) of LY3873862 | Predose up to 96 hours postdose
  PK: Tmax of LY3873862

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No